# **Informed Consent Form**

A Multicenter, Adaptive, Randomized, Blinded Controlled Trial of the Safety and Efficacy of Investigational Therapeutics for Hospitalized Patients with Acute Respiratory Distress Syndrome Associated with COVID-19

08 March 2022

NCT06729593

## Appendix A Sample Informed Consent form

**Short Title: Therapeutics for Severely III Inpatients with COVID-19 (TESICO)** 

**Sponsored by:** The University of Minnesota (UMN)/National Institute of Allergy and Infectious Diseases (NIAID)

**Funded by:** The National Heart, Lung, and Blood Institute (NHLBI) and National Institute of Allergy and Infectious Diseases (NIAID), US National Institutes of Health (NIH)

Full Title of the Study: A Multicenter, Adaptive, Randomized Blinded Controlled Trial of the Safety and Efficacy of Investigational Therapeutics for Severely III Patients with COVID-19

| SITE INVESTIGATOR: | PHONE: |
|--------------------|-----------------------------------------|
| CONSENT FOR PARTIC | IPATING IN AN NIH-FUNDED RESEARCH STUDY |

## ALL SITE INSTRUCTION THAT IS INCLUDED IN A TEXT BOX SHOULD BE REMOVED FROM THE SITE'S INFORMED CONSENT FOR PARTICIPANTS

US Office for Human Research Protections (OHRP) Requirements to be read by the sites:

PLEASE NOTE THAT THIS SAMPLE LANGUAGE DOES NOT PREEMPT OR REPLACE LOCAL IRB/EC REVIEW AND APPROVAL. INVESTIGATORS ARE REQUIRED TO PROVIDE THE LOCAL IRB/EC WITH A COPY OF THIS SAMPLE LANGUAGE ALONG WITH THE LANGUAGE INTENDED FOR LOCAL USE. LOCAL IRBs/ECs ARE REQUIRED TO WEIGH THE UNIQUE RISKS, CONSTRAINTS, AND POPULATION CONSIDERATIONS AS A CONDITION OF ANY APPROVAL. ANY DELETION OR SUBSTANTIVE CHANGE OF INFORMATION CONCERNING RISKS OR ALTERNATIVE TREATMENT MUST BE JUSTIFIED BY THE INVESTIGATOR, APPROVED BY THE LOCAL IRB/EC, AND NOTED IN THE IRB/EC MINUTES. JUSTIFICATION AND IRB/EC APPROVAL OF SUCH CHANGES MUST BE FORWARDED TO THE INTERNATIONAL COORDINATING CENTER OR COLLABORATING NETWORK. SPONSOR-APPROVED CHANGES IN THE PROTOCOL MUST BE APPROVED BY THE LOCAL IRB/EC BEFORE USE UNLESS INTENDED FOR THE ELIMINATION OF APPARENT IMMEDIATE HAZARD. NEW INFORMATION SHALL BE SHARED WITH EXISTING SUBJECTS AT NEXT ENCOUNTER, WITH ALL NEW SUBJECTS PRIOR TO INVOLVEMENT, OR AS THE LOCAL IRB/EC MAY OTHERWISE ADDITIONALLY REQUIRE.

## **Key information:**

We are asking you to join a research study about COVID-19. It is your choice whether or not you want to join. This form gives you information about the study that will help you make your choice. You can discuss this information with your doctor or family or anyone else you would like before you make your choice. Your choice will not affect the care you are getting for COVID-19.

#### What is the research question we are trying to answer?

We are studying two treatments for COVID-19. We are asking you to join the study because you are in the hospital with COVID-19 and have significant trouble with your breathing.

First, we are studying an experimental medicine, aviptadil (also called VIP), supplied by NeuroRx. We are trying to find out if giving this experimental medicine can help sick people in the hospital with COVID-19 have fewer bad effects from the disease, and if it may possibly help them get better and go home faster. We are also trying to see if it is safe.

This experimental medicine is a man-made version of a naturally occurring hormone in the body. It may decrease COVID-19 virus levels, inflammation, and blood clotting, and help protect the lung against injury. We think this experimental medicine may possibly help patients with COVID-19, and we think it will be safe, but we are not sure and so we are doing this study.

Second, we are studying a drug called remdesivir (also called Veklury) supplied by Gilead. Remdesivir is approved in the United States and many other countries for the treatment for COVID-19 in people who are in the hospital. We are trying to find out if remdesivir helps patients with your level of COVID-19 illness get better and go home faster. Remdesivir may decrease COVID-19 virus levels and lung injury. Currently we do not know if remdesivir will help people with your level of COVID-19 illness which is why we are doing this study.

#### What do you have to do if you decide to be in the study?

The study staff at your hospital will check to see if there is any reason you should not be in the study. They will check your medical history. They will look at tests commonly done for your condition. They will also check to see if you are able to get both of the drugs we are studying or just one of the drugs. For example, if you are pregnant you will not be able to receive the aviptadil or matching placebo (inactive salt solution) but you will be able to receive the remdesivir or matching placebo.

If you agree to be in the study, and you are able to get both treatments, we will assign you to one of four study groups. This will be done by random chance -- like flipping a


Aviptadil

Therapeutics for Severely III Inpatients with COVID-19 (TESICO) Master Protocol Version 3.0, 08 March 2022

coin. You will have an equal chance of getting either the active drug or placebo (salt solution) for each drug.

You will be assigned to one of the following 4 groups:



Your doctor will NOT decide and will not know which of these four options you will get. The study staff will also not know which option you will get.

If you agree to be in the study, and you are ONLY able to get Aviptadil we will assign you to one of two study groups. This will be done by random chance -- like flipping a coin. You have an equal chance of being in each group.



If you agree to be in the study, and you are ONLY able to get remdesivir we will assign you to one of two study groups. This will be done by random chance -- like flipping a coin. You have an equal chance of being in each group.



Aviptadil: You will receive the Aviptadil study product (either the experimental medicine or the matching placebo) for three consecutive days starting on the day you join the study (study Day 0). You will get it by an intravenous (IV) drip through a tube in your vein. This is called an infusion. The infusion will take about 12 hours on each day that it is given.

Aviptadil is the only thing you may be given that is experimental. It is NOT approved for use in people with COVID-19 by the United States Food and Drug Administration (FDA) or any other regulatory body in the world. It is approved in some countries outside the US for another condition but is given in a different way. Its use in the United States is strictly limited to research.

**Remdesivir:** You will receive the remdesivir study product (either the active medicine or matching placebo) once per day for up to 10 days. You will also get this by an IV drip through a tube in your vein, which will generally take 1-2 hours. Remdesivir is approved in the United States for the treatment of COVID-19 in people who are in the hospital. It's not known whether it works in people with more severe COVID-19.


**Other treatments**: As part of the study you may also get a drug called a steroid for up to 10 days while you are in the hospital, as care for your COVID-19, unless your doctor thinks the steroid would not be safe for you to take. Steroids have been shown in prior studies to help people survive COVID-19. Steroids are available for other diseases in the United States, so your doctor will be using it "off-label," which means that while there is not formal FDA approval for this use, your doctors think it is reasonable. It is likely that you would receive steroid medicine even if you were not in the study.

Any other medications or treatments you will be given will be what you would usually receive in this hospital for your condition. There may be some additional procedures or testing done for study purposes. We will describe these below.

You will be in the study for 180 days. We will check on your health every day while you are in the hospital, and regularly after you leave the hospital.

We will swab your nose to see how much of the virus that causes COVID-19 is present. We will take blood samples from you to better understand the body's response to the infection. Some of the blood may be used in future studies.

To be in the remdesivir/placebo part of the study, you will need to agree to not have sex that could make you or a partner pregnant for seven days after you finish the remdesivir or placebo infusion. This may involve not having sex at all (abstinence), or you may use effective contraception (hormonal contraception or barrier methods with spermicide) to avoid pregnancy. Methods like rhythm, sympto-thermal or withdrawal are not effective for the purpose of the study. You can ask the study team about this if you have questions or concerns.

If you are pregnant, you cannot be in the aviptadil/placebo part of the study. You can still be in the remdesivir/placebo part of the study.

If you become pregnant during the study, please let your study team know as soon as possible. We will ask to follow you until your pregnancy is over, to see if there were any problems that may have been caused by any of the study treatments.

We will need to do the following things with you, and gather detailed information at these times:



We may need to get some information from your medical record.

 By signing this consent, you agree to let us get information for this study from your medical record.

- By signing this consent, you are giving us permission to contact other hospitals
  or medical facilities if you are admitted there during the time you are in the study.
  We will contact them to be sure we know how you are doing.
- We will ask you to give us information about other people we can contact if we
  are not able to reach you after you leave the hospital, so we can find out how you
  are doing.

We will send the information we collect to the University of Minnesota (UMN) in the US where it will be stored and analyzed. In this information, only a code number, your year of birth, and a 3-letter code that the study staff chooses identifies you.

The study staff here at this site are responsible for keeping your identifying information safe from anyone who should not see it.

We will send the blood samples to a laboratory in the US for storage. We will keep them for as long as we have the funding and space to do so, which we expect to be many years. There is more information below about how we will use these samples.

#### Why would you want to be in the study?

If you get study drug, it is possible it may help you get better, or that you may get home faster, but we do not know that.

# It is important to remember that some people in this study will get inactive placebo and will not get study drug.

By being in this study, you will help doctors learn more about how to treat COVID-19 in people in the hospital. Because so many people are getting hospitalized with COVID-19, this could help others. There may be a large health impact if a treatment proves to be safe and is shown to be effective.

#### Why would you NOT want to be in the study?

Since only some people in this study will get study drug, you may not receive it. Even if you do get study drug, it may not be useful, or it may have harmful side effects, so being in the study would not be of any direct help to you.

#### What are the risks or side effects of the study treatments?

All treatments have risks and may cause side effects. These may happen to you from the study treatment.

You may have an allergic reaction, including hives, trouble breathing, or other allergic responses. Allergic reactions like these are likely to be rare, but may be severe or life-threatening.

You will be monitored very closely while you are being given the infusion of the study product (aviptadil or placebo) and for at least 2 hours after the infusion is finished. We will give you prompt medical care if needed to treat any side effects from the infusion.

There are discomforts and risks associated with blood draws. You will have these things done while you are in the hospital even if you are not in the study. These discomforts and risks are no different from what you would experience if they were performed as part of your regular hospital care for COVID-19.

#### What are the risks or side effects of Aviptadil?

One effect of aviptadil is that it relaxes smooth muscle such as in your lungs, blood vessels, and intestines. Relaxing this type of muscle opens up your airways so it is easier to breathe and get oxygen into your body.

The most common side effect of aviptadil infusion is decreased blood pressure. In early studies of very ill patients with lung injury, about 1 in 5 people (20%) had lower blood pressure during the infusion of aviptadil. The decrease was usually small and went away within 10 minutes of stopping the infusion.

Facial flushing is common with aviptadil and is not dangerous. It is caused by relaxation of the blood vessels in the skin and goes away when the infusion is stopped.

Increases in heart rate are common and usually not dangerous. The increase in heart rate is mostly due to blood vessel relaxation.

Some people getting aviptadil have had mild to moderate diarrhea. The diarrhea goes away when the infusion is stopped.

#### What are the risks or side effects of Remdesivir?

The most common side effects of remdesivir included abnormal liver function test results, abnormal blood clotting test results, constipation, diarrhea, nausea, vomiting, decreased appetite, and headache. The abnormal liver function tests lasted longer than a few days in some people but went back to normal within a few weeks or less.

Remdesivir might affect the way that other medications are processed by your body. They might stay in your body longer, or shorter, at higher or lower levels. At the time this document was written, one person in another study had an increase in the level of a medication in their blood that was considered by study doctors to be at least possibly related to having taken remdesivir. There did not appear to be any harm from this temporary change. You can ask the study team more about this if you are concerned.


Aviptadil

## Therapeutics for Severely III Inpatients with COVID-19 (TESICO) Master Protocol Version 3.0. 08 March 2022

Some people may have some side effects after the infusion of remdesivir. Other people may have no side effects.

#### What are the risks and benefits of taking steroids?

Steroids may cause your sodium (salt) and glucose (sugar) levels to rise in your blood. You may feel anxious while taking steroids. You may be given steroids to treat your COVID-19 even if you do not join this study.

#### What if you are pregnant or breastfeeding?

If you are pregnant or breastfeeding, you can still join this study, although you cannot participate in the aviptadil portion of the study. However, we do not have any information about how either aviptadil or remdesivir may affect your baby. The risks to a pregnant woman or an unborn baby might be serious. Please take this into account as you make your decision about whether to join this study.

#### Additional information:

Here is some additional information about the study that may help you make your choice about whether you want to be in the study.

The NIH, an agency of the US Federal government, is paying for this study.

We are required to comply with all rules and regulations for human research as well as the laws of each country where the study is taking place.

This study is taking place in several countries. We expect to enroll about 800 people around the world.

You do not have to join this research study if you do not want to. If you choose to join the study, you can stop at any time. If you choose not to join or to stop, the medical care you are getting now will not change.

If we get any new information that might change whether you want to join or stay in the study, we will tell you right away.

If you do not want to be in this study, you will still get the usual care to treat COVID-19. However, you cannot get Aviptadil because it is experimental.

#### What are the costs to you?

We will give you the study treatment at no cost. We will pay for all clinic visits, lab work, and other tests that are part of this study.

THE NEXT PARAGRAPH IS FOR UNITED STATES SITES ONLY. SITES IN OTHER COUNTRIES SHOULD DELETE THE NEXT PARAGRAPH.

Page o of 20

You, your insurance company, or some other third-party payer must pay for all other medicines and hospital costs.

SITES OUTSIDE THE UNITED STATES: Please replace the paragraph above with language appropriate for your location

## Will you be paid to be in the study?

We will compensate you for your time and inconvenience participating in the study. [Specific details to be completed by site.]

## What if you are hurt as part of this study?

If you are hurt because of being in this study, [insert the name of the hospital/clinic] will treat your injury right away. You or your insurance will have to pay for this treatment. The study cannot pay you or pay for any care for study-related injuries or for your illness.

If the above is not true for your site, i.e., if trial insurance covers such cost, please replace the above with appropriate language.

[The following section, up to "What happens to the blood samples?" is for US sites only.]

A Declaration under the Public Readiness and Emergency Preparedness (PREP) Act was issued by the Secretary of the United States Department of Health and Human Services on March 10, 2020. This Declaration limits the legal rights of a subject participating in clinical studies utilizing COVID-19 countermeasures. Because this study is covered by the Prep Act Declaration, covered persons, such as the manufacturers, study sponsor, researchers, healthcare providers and others have liability immunity (that is, they cannot be sued by you or your family under the laws of the United States).

If you believe that you may have been harmed as a result of this research study, certain claims for serious injury or death caused by the countermeasure may be eligible for compensation through the Countermeasures Injury Compensation Program. This is a program set up by the United States Government.

Information about this program can be found at <a href="https://www.hrsa.gov/cicp/about/index.html">https://www.hrsa.gov/cicp/about/index.html</a> or by calling 1-855-266-2427. If you are


eligible for this program, you must file a claim within one year of the administration or use of the covered countermeasure.

## What happens to the blood samples?

We will send the blood samples to a central laboratory in the United States. You and your doctor will **not** get the results of any tests done on these samples. We will not sell your samples and they will not be used for research aimed at making money (commercial research). The laboratory where the samples are stored will not have any information that could identify you.

The blood samples will measure how many COVID-19 antibodies are in your blood. This will tell us how your immune system responded to your COVID-19. The blood samples will also measure the amount of virus in your blood and other results related to your COVID infection.

Any blood samples that are left over after these tests will be stored at the central laboratory for as long as we are able to keep them. We hope to use these in the future to answer other questions about COVID-19, the virus that causes it, and how people respond to treatment. You and your doctor will **not** get any results from these tests.

You can withdraw your consent for us to keep these specimens at any time. Let your study team know if you do not want the study to keep your specimens anymore, and every effort will be made to destroy all of your specimens that are still at the central laboratory.

#### How do we protect your privacy?

We will take every reasonable step to keep your health information private and to keep anyone from misusing it.

Your information (data) and samples will not be identified by name, or in any other way, in anything published about this study.

We will do everything we can to keep your personal information private, but we cannot guarantee that nobody will get it. We may have to release your personal information if required by law.

These people may see your medical and research information:

- the [insert the name of the hospital/clinic] ethics committee (institutional review board [IRB]);
- the sponsor, the group paying for the research (US NIH), other study research staff and study monitors
- US and other participating countries' health regulatory agencies, including the US FDA.

They are committed to protecting your privacy.


As the research staff at [inset the name of the hospital/clinic], we are required to make sure that people not involved with this study cannot see your research and medical information. We will keep your research files in a safe place and will handle your personal information very carefully.

Your study data are sent electronically to the UMN in the US through a secure system. By signing this consent, you agree to having your data sent to UMN. No information that could directly identify you is sent to UMN. This is called "pseudonymized data." Access to the data at UMN is limited through security measures, and no data breach or unauthorized access has ever occurred in this system. After the study is over, the data will be stored securely for the period required by law.

Your study data will be shared with the US National Institutes of Health (which is paying for this study), and with regulators that oversee the study, including the US FDA, as required by law. Your study data will also be shared with the drug company that provides the study medicine to help them develop the drug.

UMN may share your data and specimens with other people who study COVID-19. UMN will remove any information that could possibly be used to identify you before sharing. This is called "anonymizing the data." We will not ask you for additional consent for this sharing. UMN will only share data and specimens for research projects that are approved by the group that is conducting this study.

This study has a Certificate of Confidentiality from the US Federal Government. This means that UMN cannot share any data it has about you with national, state, or local civil, criminal, administrative, legislative, or other authorities unless you specifically allow us to share it.

A description of this clinical trial will be available at http://www.ClinicalTrials.gov, and on the EudraCT website (https://eudract.ema.europa.eu/). These websites will not include your name or any other direct identifiers such as your contact information. These websites will include a summary of the results of this research once the study has been completed. You can search either website at any time.

[Note for US sites: The following brief HIPAA authorization is provided. Your sitespecific consent should be modified to reflect the HIPAA authorization language requirements at your site.]

To do this research, we will collect and use your personal data, as described above and in any HIPAA Authorization Form we have given you. Please tell us whether you agree to have us collect and use your personal data by placing your initials in front of your selection.

| Yes, I agree to the collection and processing of my personal data. |
|-------------------------------------------------------------------------|
| No, I do not agree to the collection and processing of my personal data |

**Aviptadil** 

## <u>The</u>rapeutics for <u>Severely III Inpatients with <u>COVID-19</u> (TESICO) Master Protocol Version 3.0, 08 March 2022</u>

It is your choice whether you allow us to collect and use your data. However, you will not be able to be in this study if we cannot collect and use your data.

[The following section (up to "What are your rights regarding your data?") is for **US sites** only.]

There are a lot of studies trying to find out more about COVID-19 and how people do after they have had COVID-19. Sometimes other researchers studying COVID-19 may ask if we know of people who might be interested in being in a study. If you think you might be interested in future studies, you can let us know now. We are asking you for permission to share your contact information (name, email, phone number, mailing address) with other researchers outside the study team who ask us to help them. We would only share your contact information with researchers who have appropriate ethics approval for their study. We will never share your contact information with researchers doing studies aimed at making money ("commercial research"). Even if you let us give other researchers your contact information, you do not have to be in any future studies. You always have the choice to say "no" if someone contacts you for a future study. If you tell us now that we can share your contact information but later you change your mind, let us know. If you change your mind, we will no longer share your contact information with other COVID-19 researchers.

## Please put your initials by your choice:

| <b>Yes</b> , you <b>can</b> share my contact information with other qualified researchers. |
|---|
| No, do not share my contact information with other qualified researchers. |
| It is your choice whether to let us share your contact information with other research |

It is your choice whether to let us share your contact information with other researchers studying COVID-19. You can still be in this study even if you do not want us to share your contact information.

[The following section (up to "What if you have problems or questions?") is for **only for countries subject to the GDPR or similar legislation requiring this information**. It should only be included in consents for sites subject to such legislation. It will vary from place to place whether it must be in this consent document, a separate consent document, or an information sheet that does not require signature. The amount of information provided may be reduced to meet the requirements of a particular country (e.g., not all countries/ECs require an enumeration of all of a data subject's rights).]

#### What are your rights regarding your data?

The UMN is a public research university, and this study is funded primarily by a grant from the US Federal government. UMN and the study funding source require the sponsor (UMN) to follow regulations and policies that are meant to protect your privacy. UMN is also required to comply with the General Data Protection Regulation (GDPR), because it processes data obtained from people in Europe.


There is no specific independent supervisory authority overseeing the processing of data in the US. Any complaint you might have about the use of your data would be made to your national data protection authority.

The GDPR gives you additional rights which we would like to inform you about below.

**Right to Information:** You have the right to know what data about you is being processed. You can also get a free copy of this data provided.

**Right to Correction:** You have the right to correct any information about you which is incorrect or had become incorrect.

**Right to Erasure/Anonymization:** The sponsor is required under both EU and US law to retain data from research studies like this one for many years. However, you have the right to request that your personal data be completely anonymized. This is done by destroying the information at your study center that links your identity to the pseudonymized data held by the sponsor. This means that no one would ever be able to link the data held by the sponsor to you personally.

**Right to Restriction of processing:** Under certain conditions, you have the right to demand processing restrictions, i.e. the data may then only be stored, not processed. You must apply for this. Please contact your study physician or the data protection officer of the study center if you want to do so. This right may be limited if the restriction would affect the reliability of the study results.

**Right to Data portability:** You have the right to receive the personal data that you have provided to the study center. This will allow you to request that this information be transmitted either to you or, where technically possible, to another agency designated by you.

**Right to Contradiction:** You have the right to object at any time to any specific decision or action taken to process your personal data. This right is limited for data that have already been processed and may be limited if your objection would affect the reliability of the study results.

**Right to Withdrawal of this consent:** You may withdraw your consent at any time with effect for future data collection. This withdrawal may be in an informal or verbal communication to your investigator. If you withdraw your consent this will not affect the lawfulness of the data processing that has been or will be done with data collected until you withdraw consent. Data already collected will be anonymized.

If you would like to use one of these rights, please first contact the person responsible for the data collection at your study center:

| Person responsible for data collection at the study center: |
|-------------------------------------------------------------|
| Name: |
| Address: |
| Phone: |
| Email |

For concerns about data processing and compliance with data protection requirements you can also contact the data protection officer responsible for the study center:

| Data protection officer responsible for the study center: |
|-----------------------------------------------------------|
| Name: |
| Address: |
| Phone: |
| Email |

In addition, you have the right to lodge a complaint with the competent authority if you believe that the processing of personal data concerning you is contrary to the GDPR:

# Data protection authority responsible for the study center: Name: Address: Phone: Email

#### What if you have problems or questions?

If you ever have questions about this study, or about the storage or use of your data or samples, or if you are hurt by being in the study, contact:

- [name of the investigator or other study staff]
- [telephone number of the above]

If you have questions about your rights as a research participant, you can call:

- [name or title of person on the ethics committee (IRB) or other organization appropriate for the site]
- [telephone number of the above]

#### SIGNATURE PAGE FOR CONSENT TO PARTICIPATE IN THE TESICO STUDY

I have read the consent or have had it explained to me. I believe that I understand the information. By signing and dating this consent, I am stating that I want to join this study. I understand that I do not waive any of my legal rights as a study participant by signing this consent. I understand that I will receive a copy of the signed and dated consent.

| If you agree to be in this study, please sign below. | |
|------------------------------------------------------|-------|
| | Date: |
| Signature of participant | |
| Printed name of participant | |
| | Date: |
| Signature of investigator/designee | |
| Printed name of investigator/designee | |
| FOR ADULTS NOT CAPABLE of GIVING CONSENT | |
| | Date: |
| Signature of Legally Authorized Representative (LAR) | |
| Printed name of LAR | |

| <u>The</u> rapeutics for <u>Severely III Inpatients with <u>COVID-19</u> (TESICO) Master Protocol Version 3.0, 08 March 2022</u> | |
|---|---|
| Relationship of LAR to Participant | |
| (Indicate why the LAR is authorized to act as a surrogate health care decision-make<br>under state or applicable local law) | r |

#### Witness to Consent Interview

On the date given next to my signature, I witnessed the consent interview for the research study named above in this document. I attest that the information in this consent form was explained to the subject, and the subject indicated that his/her questions and concerns were adequately addressed.

| | Date: |
|-------------------------|-------|
| Signature of witness | |
| Printed name of witness | |

NOTE: This consent form, with the original signatures, MUST be retained on file by the Investigator of Record. A copy of the signed and dated consent must be given to the participant. A copy should be placed in the participant's medical record, if applicable.

If no-touch / electronic consent is used, the participant must be provided with a copy of the consent in a manner appropriate to the method used to obtain it. A record of the act of consent must also be appropriately retained in the participant's medical record.

Therapeutics for Severely III Inpatients with COVID-19 (TESICO) Master Protocol Version 3.0. 08 March 2022

#### <u>Additional Consent for Genetic Testing on Stored Specimens</u>

WHY IS GENETIC TESTING BEING DONE? The study team would like your permission to collect a small amount of your blood and store them for researchers who will do genetic testing (testing on your genes) and other related tests in the future. These tests will help us understand how the genetic makeup of people affects the COVID-19 virus and how it makes people sick.

Any future research done on the blood collected for this study will be related to the COVID-19 virus for which you are being studied in this trial.

#### WHAT WILL HAPPEN DURING GENETIC TESTING?



If you agree to take part in this study, three blood specimens will be collected along with other blood being drawn for the study, approximately 15 mL (about 1 tablespoon) in total. The blood will be taken with other laboratory test samples so you will not get an extra needle stick.

HOW WILL YOUR BLOOD BE USED? Your blood will be used to learn more about the health problems that may be caused by COVID-19. This may include tests to better understand why some people have more severe complications (get sicker) than others and why medicines to prevent or treat these infections might work better in some people than in others.

Researchers involved with this blood collection project do not know yet exactly which tests will be done.

You and your study doctor or nurse will not get any results from the tests done on your blood collected for this genomics study. These tests will only be used for research and may not apply to your medical care.

Your blood sample collected for this study will:

- Become the property of INSIGHT.
- Not be sold or used to make commercial products.
- Not be tested for any specific research study unless the plan for using your blood is approved - based on scientific and ethical considerations - by the INSIGHT Scientific Steering Committee, the U.S. National Institutes of Health (NIH), and a special committee (an Institutional Review Board or Ethics Committee) at the researcher's institution.

## HOW WILL YOUR PRIVACY AND THE CONFIDENTIALITY OF YOUR **INFORMATION BE PROTECTED?**


Every reasonable step will be taken to protect your privacy and the confidentiality of your health information and to prevent misuse of this information, and to make sure your blood sample is handled with care at the storage facility. For example, your research records will be identified only by a code. Your blood sample and results of any genetic testing will be identified by a second code. Only a few statisticians (persons who analyze the study results) associated with the INSIGHT studies will have access to both codes in order to analyze the test results. These statisticians will not have access to any information that can identify you.

Researchers will write reports, including information they learn from future tests on your blood. These reports will be shared with participating research sites. These findings will also be submitted for publication in scientific or medical journals. When the results of the research are published or discussed in conferences, no information will be included that would reveal your identity.

However your records may be seen by:

- Institutional Review Boards (IRBs) or Ethic Committees (ECs) who review the study to make sure it is ethically acceptable
- Agencies of the U.S. government that fund or oversee this research, for example, the U.S. National Institutes of Health (NIH) or the U.S. Office for Human Research Protections (OHRP)
- Research staff and study monitors, and their designees.

Staff at **[insert the name of the site]** will handle your personal information very carefully. They are required to make sure that people not involved with this study do not have access to your research and medical records.

## [For U.S. Sites Only]

In addition to these efforts to keep your information confidential, the INSIGHT Genomics study is covered by a *Certificate of Confidentiality* from the U.S. Department of Health and Human Services. This certificate means that researchers cannot be forced to give information collected as part of this study to people who are not involved with the study, for example, the court system. However, this certificate has limited protection rights. You should know that it does not stop the doctor in charge of this study from taking appropriate steps to prevent serious harm to yourself or others. Federal and state laws also help protect research participants and others who have genetic testing done.

## [For International Sites Only]

Efforts will be made to keep your personal information confidential, but we cannot guarantee complete confidentiality. Your personal information may be released if


required by law. Any publication of this study will not use your name or identify you personally.

#### HOW LONG WILL YOUR BLOOD BE KEPT?

Your blood specimen will be stored as long as funding is available for storage and testing.

## [Alternative to Previous Paragraph for non-US Sites Only]

Your blood specimen will be stored safely and securely at a special facility called a specimen repository. The repository may be located in the United States. This facility follows strict procedures so that only approved researchers can use the stored specimen for future testing. The employees at this facility who will store and track your blood specimen will not have information that identifies you by name.

**Risks:** There are few risks involved with your participation in this study. Having your blood drawn may result in a little pain and slight bruising where the needle goes into your skin. You may also feel lightheaded, bleed, develop a small blood clot where the needle goes into your skin, or faint. Very rarely, your skin may get infected. Another small but unlikely risk is the possibility of others finding out about your participation in this study.

**Benefits:** You will not receive any direct benefit from your samples. Information obtained from the tests may provide useful information, to help other patients, about the causes, risks, and prevention of the COVID-19 virus.

WHAT IF YOU DON'T WANT YOUR BLOOD FOR GENETIC TESTING STORED ANY LONGER? If you sign the consent that your blood can be stored for research to be done at a later date you can change your mind at any time. If you change your mind, you must write a letter to [insert the name of the principal investigator] at the [insert the name and address of the site] to let them know that you do not want your blood specimen collected for this study used for future research. A sample letter will be given to you as a guide to help you express your request in writing.

When *[insert the name of the principal investigator]* receives your letter, the research staff will contact you to come to the clinic to verify your decision by signing and dating this original informed consent form. A second copy of this consent will be given to you as proof that we received your request. If we do not hear from you within 30 days after getting your letter to withdraw from this study, we will send your request to the storage facility.

If you decide to withdraw consent for this study, your blood sample, including any parts separated from the sample, will not be used. Every effort will be made to destroy your


blood sample and any parts separated from it. If some testing has already been done on your blood sample, the results from this testing will remain as part of this research. The research staff at the *[insert the name of the site]* will notify you of the date your blood specimen and any of its parts were destroyed.

**Costs or compensation of study:** There will be no costs to you or compensation.

**Consent:** Please *mark the box for* yes or no and *sign your name*, indicating you have freely given your answers and consent:

| My blood samples may be stored and used for future genetic research | |
|---------------------------------------------------------------------|------|
| in COVID-19 or other serious illness: | No □ |
| Signature (subject or surrogate) Date | _ |
| Subject or Surrogate Printed Name | |
| Signature of Person Obtaining Consent Date | _ |
| Printed Name and Title of Person | |